CLINICAL TRIAL: NCT03237754
Title: Clinical and Neuronal Changes in Chronic and Episodic Migraine Patients After Neurostimulation
Brief Title: Neurostimulation in Chronic and Episodic Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems (especially for chronic migraine patients)
Sponsor: University of Zurich (Other)
Collaborators: Kantonsspital Baden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2016-00646
Record Dates: First submitted 2017-07-28; First posted 2017-08-03 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Double-blind Design; Sham-controlled; Randomized
Keywords: migraine; neurostimulation; neuroimaging; tDCS; MRI
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: Patients receive either Placebo or real neurostimulation
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Neurostimulation (Experimental): 4 weeks of neurostimulation (using tDCS)
  Interventions: Device: tDCS device from neuroConn
- Sham Neurostimulation (Sham Comparator): 4 weeks of sham Treatment with the same device used for real neurostimulation
  Interventions: Device: tDCS device from neuroConn

INTERVENTIONS:
Device: tDCS device from neuroConn — weak electrical direct current stimulation

SUMMARY:
Currently, successful prevention of migraine is not sufficiently achieved by (prophylactic) drug therapy. In contrast, neurophysiologically guided treatments might provide an alternative avenue, since these can normalize brain alterations without side effects. Transcranial direct current stimulation (tDCS) appears useful in the acute and prophylactic treatment of migraine, probably because of its modifying and re-balancing influence on neuronal activity. Yet, to test for the efficacy of tDCS in a clinically acceptable way, it is necessary to apply not only tDCS but also a "sham" placebo, which is often neglected in tDCS stimulation studies. Further, tDCS needs to be applied in a large (n > 20) sample of well-defined migraine patients, which would be advantageous, compared to previously published work. Monitoring sources of regional neuronal alterations in migraineurs prior and after tDCS is essential to investigate physiological mechanisms of tDCS. There is an increasing interest towards non-pharmacological treatment alternatives for migraine (and headache disorders) with reduced side effects to established prophylactic medications. The primary outcome of this project is to demonstrate that repetitive sessions of neurostimulation lead to a significant and permanent reduction of the primary symptom severity (i.e. migraine attacks) for patients suffering from chronic and episodic migraine. Since neurostimulation tools are nowadays accepted as therapeutic tools, our study might provide evidence that tDCS can be a non-pharmacological alternative for treating migraine.

ELIGIBILITY:
Inclusion Criteria:

Patients from age 18 upwards (max. 80 years) suffering from chronic or episodic migraine. Medication overuse headache (MOH) patients are included as well (as chronic migraine patients do often show MOH).

Healthy volunteers (18-80 years) are included if they don't fulfil the exclusion criteria and do not suffer from migraine or other headache disorders, except infrequent episodic tension-type headache All volunteers are able to read and sign the informed consent.

Exclusion Criteria:

Patients and healthy volunteers are excluded if they fulfil one of the following exclusion criteria:

Common MR exclusion criteria: such as metallic items in the body (i.e. eye splinter, MR incompatible implants*), pacemaker, claustrophobia or obesity (body mass index > 35).

Also pregnant participants and participants suffering from a degenerative disorder of the Central Nervous System, such as Stroke, Multiple Sclerosis, Parkinson's Disease, Alzheimer's Disease and Huntington's Disease will be excluded. Participants with major psychiatric disorders such as schizophrenia, bipolar disorder will also be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Migraine days | 6 months
  Change in migraine days (in episodic and chronic migraine patients) after tDCS Treatment (relative to before tDCS)Treatment) in the active and Placebo group

SECONDARY OUTCOMES:
MR data | 6 months
  Changes in functional and structural MR data before and after tDCS Treatment
Clinical data | 6 months
  Clinical variables (e.g. depression scores) will be compared in an identical fashion as for the variable "migraine days

CONTACTS AND LOCATIONS:
Overall Officials: Lars Michels, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pohl H, Sandor PS, Moisa M, Ruff CC, Schoenen J, Luechinger R, O'Gorman R, Riederer F, Gantenbein AR, Michels L. Occipital transcranial direct current stimulation in episodic migraine patients: effect on cerebral perfusion. Sci Rep. 2023 Aug 25;13(1):13944. doi: 10.1038/s41598-023-39659-5. PMID 37626074
- [Derived] Schading S, Pohl H, Gantenbein A, Luechinger R, Sandor P, Riederer F, Freund P, Michels L. Tracking tDCS induced grey matter changes in episodic migraine: a randomized controlled trial. J Headache Pain. 2021 Nov 20;22(1):139. doi: 10.1186/s10194-021-01347-y. PMID 34800989